CLINICAL TRIAL: NCT04750265
Title: Robotic Assisted Early Mobilization in Ventilated ICU Patients With COVID-19: an Interventional Randomized, Controlled Feasibility Study (ROBEM II Study)
Brief Title: Robotic Assisted Early Mobilization in Ventilated ICU Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Reactive Robotics GmbH (Unknown)
Responsible Party: Principal Investigator, Stefan J Schaller, Deputy Clinical Director, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROBEM II
Record Dates: First submitted 2021-02-09; First posted 2021-02-11 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Covid19; Critical Illness; Critical Illness Polyneuromyopathy; Early Mobilization; Rehabilitation; Robotics
Keywords: COVID19; Early mobilization; robotics; Vemo
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel-group, open label pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic assisted early mobilization (Experimental): Early mobilization therapy assisted with robotics
  Interventions: Device: Robotic assisted early mobilization
- Standard Care (No Intervention): Mobilization according to standard care by staff

INTERVENTIONS:
Device: Robotic assisted early mobilization — Robotic assisted early mobilization Robotic assisted early mobilization started within 72 hours of ICU admission.
  Arms: Robotic assisted early mobilization

SUMMARY:
Feasibility trial investigating the potential higher frequency of robotic assisted early mobilization in intubated COVID19 patients on the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Invasive mechanically ventilated and expected to be ventilated for another 24 hours
* Cardiovascular stability, allowing mobilization
* Respiratory stability, allowing mobilization

Exclusion Criteria:

* Bed-bound before ICU admission
* Bed-rest order or contraindication of weight load of the lower extremity or spine
* Severe skin lesions or fasciitis in the area of contact with the device or rhabdomyolysis
* Fresh SAB, ICB or elevated ICP
* Status epilepticus
* Acute intoxication
* Shock with catecholamine doses >0.3μg/kg/min or acute bleeding including organ ruptures
* Multiorgan failure with lactate > 4 mmol/l
* Body height outside the range 150-195 cm
* Body weight outside the range 45-135 kg
* pAVK IV°
* Pacemakers or other electrical stimulators
* Implanted medical pumps
* Pregnancy
* Life expectancy below 7 days or acute palliative care situation
* Death inevitable or maximum therapy is not carried out by the treating physicians or due to patient's request
* Unable to understand the official language

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Level of mobilization | 5 days
  Level of mobilization during the first 5 days after admission on the ICU, measured with the ICU-Mobility Scale (0-10)
Level of mobilization | 5 days
  Level of mobilization during the first 5 days after admission on the ICU, measured with the Surgical Optimal Mobilization Scale (0-4)

SECONDARY OUTCOMES:
Frequency of Mobilization | 5 days
  Frequency of early mobilization during mechanical ventilation
Initiation of first Mobilization | 5 days
  Time of first mobilization after admission on ICU (in hours)
Mobilization duration | 5 days
  Average duration of mobilization sessions during mechanical ventilation (in min)
Depth of sedation | 5 days
  Depth of sedation measured with RASS during the first 5 days after admission on ICU
Days of sedation | during ICU stay (normally up to 30 days)
  Days under sedative medication during ICU stay
Days of mechanical ventilation | during ICU stay (normally up to 30 days)
  Days of mechanical ventilation during ICU stay
Days of Intubation | during ICU stay (normally up to 30 days)
  Days of Intubation during ICU stay
Days of Delirium | during ICU stay (normally up to 30 days)
  Days of Delirium during ICU stay
MRC Score | One time point before ICU Discharge
  MRC Score at ICU Discharge
Muscle wasting | 5 days
  Muscle wasting assessed using ultrasound measurement of the M. femoris
Number of Health care provider | 5 days
  Number of Health care provider needed for mobilization
Mortality | at 180 days after study start
  Mortality during ICU and Hospital stay and 180 days after admission at ICU
Length of stay | Hospital stay (approx. 30 days)
  Length of stay at ICU , in Hospital (in days)
Global function | at 180 days after study start
  Global function measured with WHODAS
Health care provider assessment | 5 days
  Assessment of the satisfaction with the mobilization by the health care provider using Likert-Scales (1-5)
Safety events | 5 days after study start
  Frequency of safety events during mobilization
Functional status | at 180 days after study start
  Measurement of ADLs/IADLs for which patients need assistance
DRG workplace data | Hospital stay (approx. 30 days)
  expenses of the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Univiversitätsmedizin Berlin, Mitte, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Depersonalized data can be requested from the PI after publication of the study for scientific purpose.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publishing results.
Access Criteria: Data will be shared to other researchers on reasonable request.